CLINICAL TRIAL: NCT01925573
Title: Proposed Pilot Study of Combined Optune+ Bevacizumab, and Hypofractionated Stereotactic Irradiation for Bevacizumab-Naive Recurrent Glioblastoma
Brief Title: Optune(NOVOTTF-100A)+ Bevacizumab+ Hypofractionated Stereotactic Irradiation Bevacizumab-Naive Recurrent Glioblastoma (GCC 1344)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00056719
Record Dates: First submitted 2013-08-13; First posted 2013-08-19 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: RECURRENT GLIOBLASTOMA; Brain Tumor
Keywords: RECURRENT GLIOBLASTOMA; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Optune+RT+Bevacuzimab (Other): Part 1:
  Bevacizumab every 2 weeks plus Optune daily for 4 week cycles.
  Part 2:
  RT will begin post 3 round of Bevacizumab (hypofractionated radiotherapy: 30 Gy in 5 fractions or 35 Gy in 10 fractions) per physician choice.
  Part 3:
  Adjuvant Bevacizumab and Optune
  Interventions: Device: Optune(NOVOTTF-100A)

INTERVENTIONS:
Device: Optune(NOVOTTF-100A)

SUMMARY:
This protocol is designed to generate and provide preliminary data to determine the safety and activity of combination therapy using tumor treating fields (TTFields; Optune(NovoTTF-100A); Novocure, Haifa, Israel), a novel FDA-approved therapy utilizing alternating electric fields to inhibit tumor cell growth, along with bevacizumab (Avastin; Genentech, San Francisco, CA), a humanized monoclonal antibody that inhibits vascular endothelial growth factor (VEGF), and hypofractionated stereotactic radiotherapy, a highly-focal abbreviated course of brain irradiation, in the treatment of patients with bevacizumab-naive recurrent GBM. Each of these individual therapies, and also several combinations in doublets, has already demonstrated safety and efficacy but prospective clinical data for the concurrent combination of all three therapies are lacking.

DETAILED DESCRIPTION:
The combination of Optune(NovoTTF) with the active regimen of bevacizumab and hypofractionated stereotactic radiotherapy bases the addition of an effective new treatment in the setting of a safe regimen with favorable survival reports. To date, no clinical data are available on the interaction of concomitant tumor treating fields with radiation therapy either with or without bevacizumab. TTF and radiation both have the potential to enhance the other's therapeutic ratio though synergistic mechanisms of action. The addition of bevacizumab to this regimen has both therapeutic and improved-toxicity implications. A trial combining Optune with the proven regimen of HFSRT and bevacizumab for recurrent glioblastoma affords an avenue to demonstrate safety in a population who may more readily derive a benefit from novel multimodality therapy and explore the potential for synergistic effect. The endpoint of efficacy would clearly need to be more definitively addressed in a future categorical trial, which would be the logical positive outcome of this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* 1 Patients with recurrent or progressive glioblastoma or other grade IV malignant glioma (i.e. glioblastoma, gliosarcoma, giant cell glioblastoma, etc.) who have failed prior radiation but who have not progressed/recurred on bevacizumab. Patients will be eligible if the original histology was lower-grade glioma and subsequent diagnosis of glioblastoma or gliosarcoma is made.

  2 Patients with any number of recurrences are allowed. 3 Brain MRI demonstrates an enhancing tumor < 8 cm in largest diameter. 4 Karnofsky performance status ≥ 70%. 5 Age ≥ 22 years old. 6 Patients must have the following laboratory values:
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin (Hgb) > 10 g/dL
  * Serum total bilirubin: ≤ 1.5 x ULN
  * ALT and AST ≤ 3.0 x ULN
  * Adequate Renal Function: BUN and Cr < 2.0 x ULN
  * Blood coagulation parameters: international normalized ratio (INR) ≤ 1.5 for patients not on warfarin 7 Minimum interval since completion of radiation treatment is 12 weeks. 8 History of standard dose CNS radiotherapy: radiation of 60 Gy in 30 fractions or 59.4 Gy in 1.8 Gy fractions, or equivalent or lower doses.

    9 Minimum interval since last major surgery, open biopsy, or significant traumatic injury is 4 weeks 10 Minimum interval since last drug therapy:
  * 3 weeks since last non-cytotoxic therapy
  * 3 weeks must have elapsed since the completion of a non-nitrosourea-containing chemotherapy regimen
  * 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen. 11 Patients must have signed an approved informed consent and authorization permitting release of personal health information.

    12 Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Female patients of child-bearing potential must have a negative pregnancy test.

    13 Patients with history of prior invasive malignancy (except non-melanomatous skin cancer) must have been disease free for a minimum of 1 year.

    14 Patients must be maintained on a stable corticosteroid regimen from the time of their baseline scan until the start of treatment and/or for at least 5 days before starting treatment.

    15 Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria: 16 No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices) 17 In-range INR (max ≤ 3) on a stable dose of oral anticoagulant for greater than 1 month or on a stable dose of low molecular weight heparin

Exclusion Criteria:

* 1 Any prior therapy with bevacizumab 2 Any significant hemorrhage defined as > 1 cm diameter of blood seen on the MRI or CT scan. If > 1 cm of acute blood is detected, the patient will be ineligible for this trial.

  3 Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury.

  4 Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:
  * History or presence of serious uncontrolled ventricular arrhythmias
  * Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE)
  * Uncontrolled hypertension (defined by a SBP ≥ 160 mm Hg or DBP ≥ 100 mm Hg while on anti-hypertensive medications) or history of hypertensive crisis or hypertensive encephalopathy, stroke, TIA, symptomatic peripheral vascular disease, or grade 2 CHF 5 Patients with cirrhosis, or active viral or non-viral hepatitis. 6 Patients with peptic ulcer, abdominal fistula, gastrointestinal perforation, intra-abdominal abscess within 6 months of enrollment.

    7 Implanted pacemaker, defibrillator or deep brain stimulator, other implanted electronic devices in the brain or documented clinically significant arrhythmias.

    8 Infra-tentorial tumor. 9 Known sensitivity to conductive hydrogels. 10 Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory).

    11 Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol 12 Pregnant or breast-feeding women. 13 Patients unwilling or unable to comply with the protocol. 14 Patients treated on any other therapeutic clinical protocols within 3 weeks of starting on this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Young, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Optune+RT+Bevacuzimab: Part 1:
  Bevacizumab every 2 weeks plus Optune daily for 4 week cycles.
  Part 2:
  RT will begin post 3 round of Bevacizumab (hypofractionated radiotherapy: 30 Gy in 5 fractions or 35 Gy in 10 fractions) per physician choice.
  Part 3:
  Adjuvant Bevacizumab and Optune
  Optune(NOVOTTF-100A)
Period: Overall Study
Arm/Group | Optune+RT+Bevacuzimab
Started | 7
Completed | 0
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Optune+RT+Bevacuzimab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.7 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5
  African American | 1
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Grade 3 or High Toxicity/Adverse Event (Primary Measure)
Description: The ability to complete protocol treatment (i.e. tri-modality treatment) without undue acute toxicity as defined below
  * : <40% rate of Grade 3 or higher nonhematologic toxicity.
  * : <15% rate of Grade 4 or higher nonhematologic toxicity
  * : <5% rate of Grade 4+ scalp dermatitis
  * : <50% rate of Grade 2-3 scalp dermatitis
  Early stopping rules: Two or more Grade 2 or higher symptomatic CNS hemorrhages; Eight treatment-related Grade 3 or higher non hematologic or Grade 4 or higher hematologic toxicities.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optune+RT+Bevacuzimab
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: AEs were evaluated per protocol during radiation and chemo, as well as during the follow-up period. Radiation and concurrent chemo lasted 6-7 weeks. Adjuvant chemo lasted 6-12 months after completion of radiation.
Description: Systematic assessment was done through regular physician assessments.
Arm/Group | Optune+RT+Bevacuzimab
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optune+RT+Bevacuzimab (N=7)
Hypertension (Vascular disorders) | 2
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Cranial- CN II Vision (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optune+RT+Bevacuzimab (N=7)
Tinnitus (Ear and labyrinth disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Hypertension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 1
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Edema: limb (General disorders) | 1
Alkaline phosphatase (Investigations) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Creatinine (Investigations) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Facial (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Left-sided (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Right-sided (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Mental status (Nervous system disorders) | 2
Mental status (Nervous system disorders) | 1
Mood alteration - Agitation (Psychiatric disorders) | 2
Mood alteration - Anxiety (Psychiatric disorders) | 3
Mood alteration - Anxiety (Psychiatric disorders) | 1
Mood alteration - Depression (Psychiatric disorders) | 2
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Flu-like syndrome (General disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated due to poor accrual. No analysis was done due to having not met accrual for study analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT01925573/Prot_SAP_000.pdf